CLINICAL TRIAL: NCT02047851
Title: Randomized, Blinded, Sham-controlled Trial of Acupuncture for the Management of Joint Pain in Patients With Psoriasis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough study participants, difficulties in recruitment
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: Aage Bangs Fond (Other)
Responsible Party: Principal Investigator, Annesofie Faurschou, MD, PhD, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-1-2013-122
Record Dates: First submitted 2014-01-26; First posted 2014-01-28 (Estimated); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Psoriasis; Arthralgia
MeSH Terms: conditions — Psoriasis; Arthralgia | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Acupuncture in active points (Active Comparator): Patients in this group will receive real acupuncture
  Interventions: Other: Acupuncture
- Acupuncture in non-active points (Sham Comparator): Patients in this group will receive acupuncture, but in non-active points
  Interventions: Other: Acupuncture
- No treatment, just observation (No Intervention): Patients in this group will receive no treatment and will only be observed.

INTERVENTIONS:
Other: Acupuncture — Patients are randomized to real acupuncture or sham acupuncture if they are in the intervention group
  Arms: Acupuncture in active points; Acupuncture in non-active points

SUMMARY:
The purpose of this study is to determine whether acupuncture is helpful for patients with joint pain associated with psoriasis

DETAILED DESCRIPTION:
In this study, patients with psoriasis and joint pain will receive either real acupuncture or sham acupuncture to see if acupuncture can be an effective treatment of joint pain in patients with psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Plaque psoriasis
* Pain from at least two peripheral joints and/or inflammatory back pain
* No or stabile treatment of the psoriasis the last 3 months
* No or stabile pain treatment the last 3 months
* Oral and written information given
* Written consent signed

Exclusion Criteria:

* Arthritis with Ultrasound verified intra articular fluid og clinical verified joint swelling
* Pregnancy og breastfeeding
* Previous treatments with acupuncture
* Treatment with anticoagulants (vitamin K-antagonists, low molecular weight heparin, unfractionated heparin, direct thrombin inhibitors, direct factor Xa inhibitors)
* Unwilling to follow protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-10; Primary Completion 2018-05-09 (Actual); Study Completion 2018-05-09 (Actual)

PRIMARY OUTCOMES:
Pain measured on the VAS | From day 0 to day 60 of the trial
  Patients will record their level of pain in a journal each day, ranging from 0 to 10 where 0 is no pain and 10 is worst possible pain.
Improvement in life quality measured with the DLQI (Dermatology Life Quality Index) | From day 0 to day 60 of the study period
  On day 0, 30 and 60 the patients will fill out a simple questionnaire with 10 questions concerning their life quality

SECONDARY OUTCOMES:
Approvement in skin lesions | From day 0 to day 60 of the study period
  At each of the 3 control visits the patients will be asked if their psoriatic skin lesions have become better from the acupuncture, and if they say yes, how much better? Minimal improvement, moderate improvement og big improvement?

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Gentofte University hospital, Hellerup
  - The departement of allergy and dermatology, Gentofte Hospital, Hellerup